CLINICAL TRIAL: NCT01742585
Title: ASP1585 Phase 3 Randomized Double Blind Placebo-controlled Study in Chronic Kidney Disease (CKD) Patients With Hyperphosphatemia Not on Dialysis
Brief Title: A Phase 3 Study of ASP1585 in Chronic Kidney Disease Patients With Hyperphosphatemia Not on Dialysis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1585-CL-0101
Record Dates: First submitted 2012-12-04; First posted 2012-12-05 (Estimated); Last update posted 2014-07-16 (Estimated); Status verified 2014-07

CONDITIONS: Chronic Kidney Disease; Renal Insufficiency; Hyperphosphatemia
Keywords: CKD; Not on dialysis; ASP1585; Bixalomer
MeSH Terms: conditions — Renal Insufficiency, Chronic; Renal Insufficiency; Hyperphosphatemia | interventions — bixalomer

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- ASP1585 group (Experimental)
  Interventions: Drug: ASP1585
- placebo group (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: ASP1585 — oral
  Other Names: LY101; AMG223; bixalomer
  Arms: ASP1585 group
Drug: placebo — oral
  Arms: placebo group

SUMMARY:
This is a randomized, double blind, placebo-controlled multi-center study to examine the efficacy and safety of ASP1585 in chronic kidney disease patients with hyperphosphatemia not on dialysis.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients (eGFR < 60 mL/min/1.73 m2)
* Serum phosphorus measurement ≧4.6 mg/dl, <9.0 mg/dl
* Written informed consent

Exclusion Criteria:

* Patients with gastrointestinal surgery or enterectomy
* Patients with severe cardiac diseases
* Patients with severe constipation or diarrhea
* Patients with a history or complication of malignant tumors
* Patients with uncontrolled hypertension
* Patients treated with parathyroid intervention within 6 months

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-10; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Change from baseline in serum phosphorus level at the end of treatment | Baseline and Week 12 or treatment discontinuation

SECONDARY OUTCOMES:
Achievement rate of the target range of serum phosphorus level | During 12 week treatment
Time to achieve the target range of serum phosphorus level | During 12 week treatment
Time-course changes in serum phosphorus levels | During 12 week treatment
Time-course changes in serum calcium levels | During 12 week treatment
Safety assessed by the incidence of adverse events, vital signs, labo-tests and 12-lead ECGs | During 12 week treatment

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Astellas Pharma Inc
Locations (5):
- Japan (5):
  - Chūbu
  - Hokkaido
  - Kansai
  - Kanto
  - Kyushu

REFERENCES:
- [Derived] Natale P, Green SC, Ruospo M, Craig JC, Vecchio M, Elder GJ, Strippoli GF. Phosphate binders for preventing and treating chronic kidney disease-mineral and bone disorder (CKD-MBD). Cochrane Database Syst Rev. 2025 Jun 27;6(6):CD006023. doi: 10.1002/14651858.CD006023.pub4. PMID 40576086